CLINICAL TRIAL: NCT02714946
Title: Prospective Randomized Comparative Study of the Effectiveness and Safety of Ultrasound-guided Laser and Radiofrequency Ablation for the Treatment of Benign Thyroid Nodules
Brief Title: Laser Ablation Versus Radiofrequency Ablation for Thyroid Nodules
Acronym: LARA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Dr. Silvia Manfrini, Medical Doctor, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Studio 96-15 CE 93321
Record Dates: First submitted 2016-02-19; First posted 2016-03-22 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Thyroid Nodule
Keywords: Thyroid Nodule; Percutaneous radiofrequency ablation (RFA); Percutaneous laser ablation (LA)
MeSH Terms: conditions — Thyroid Nodule | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LA Arm (Active Comparator): Percutaneous Laser Ablation
  Interventions: Device: Percutaneous Laser Ablation
- RFA Arm (Active Comparator): Percutaneous Radiofrequency Ablation
  Interventions: Device: Percutaneous Radiofrequency Ablation

INTERVENTIONS:
Device: Percutaneous Laser Ablation — Single session with standardized approach: One or two fibers will be used for treatments including one to three illuminations with a fixed output power of 3 W, using the pullback technique. Energy for each emission will be 1200-1800J based on nodule volume. The treatment is performed under local anesthesia and conscious sedation.
  Arms: LA Arm
Device: Percutaneous Radiofrequency Ablation — Single session with standardized approach: A radiofrequency generator and a 17-gauge, 15-cm electrode with a 1-cm active tip will be used. A transisthmic approach along the short axis of the nodule will be used and the nodules will be managed with the moving-shot technique. 60 W of radiofrequency outpower will be used for all nodules. The treatment is performed under local anesthesia and conscious sedation
  Arms: RFA Arm

SUMMARY:
The purpose of this study is to prospectively compare percutaneous radiofrequency ablation (RFA) versus percutaneous laser ablation (LA) for the treatment of solid thyroid nodules.

DETAILED DESCRIPTION:
Nodular thyroid disease is a common clinical problem whose prevalence increases with age and with a more widespread use of thyroid ultrasonography. Although most thyroid nodules are benign and need only periodic monitoring, some may require treatment for associated pressure and/or cosmetic symptoms. Although thyroid surgery is the main therapeutic approach for compressive thyroid nodules, it may be associated with several drawbacks. Long-term levothyroxine suppression treatment in elderly patients with large nodular goiters is unsatisfactory because it is ineffective. Furthermore, it is associated with adverse effects on bones and the cardiovascular system. Nonsurgical, minimally invasive treatment modalities such as percutaneous laser ablation (LA) and radiofrequency ablation (RFA) have been used to treat thyroid nodules. However no studies comparing LA and RFA have been published so far.

Aims of the study

1. To evaluate whether LA and RFA cause a reduction ≥50% in the volume of thyroid nodules after 6 months and 1 year follow-up
2. To evaluate whether the features of thyroid nodules as evaluated by thyroid ultrasound, contrast-enhanced ultrasound, power-doppler and core-biopsy influence LA and RFA outcomes
3. To evaluate changes in thyroid function and thyroid autoimmunity after LA and RFA.
4. To evaluate differences between LA and RFA in terms of complications, side effects and tolerability.

Patients will be recruited, treated and followed at Santa Maria Goretti Hospital in Latina, Italy, by physicians with expertise in LA and RFA. The scientific coordinator of this study is dr. Silvia Manfrini.

ELIGIBILITY:
Inclusion Criteria:

* Solitary thyroid nodule or dominating nodule which is well-identifiable in multinodular goiter.
* Compressive and /or cosmetic symptoms caused by thyroid nodule or increase in nodule volume >20% in 1 year even without symptoms
* A nodule volume ≥ 5 ml
* Solid nodule (uniformly compact or nearly completely solid, with a liquid component not exceeding 30%);
* Two thyroid biopsies resulted negative for malignancy
* Calcitonin levels within normal ranges

Exclusion Criteria:

* Hyperfunctioning lesion as evaluated biochemically and/or by 99mTc scintigraphy
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of thyroid nodules with volume reduction at 6 and 12 months after treatment | 12 months
  Differences in the percentage of nodules with greater than 50% base volume reduction at 6 and 12 months

SECONDARY OUTCOMES:
Basal Volume of Thyroid Nodules as Predictive factor of response to treatment | 12 months
  Basal volume in mL of the nodules will be calculated with the ellipsoid formula
Histopathological features of Thyroid Nodules as Predictive factor of response to treatment | 12 months
  % of amount of fibrosis and colloid components evaluated with score-biopsy
Variation in TSH levels after treatment | 12 months
  Variation in TSH value (mUI/ml) before and after LA and RFA
Variation in AbTPO and AbTg levels after treatment | 12 months
  Variation in AbTPO and AbTg levels (UI/ml) before and after LA and RFA
Complications | Up to 1 year follow-up
  Differences in the rate of complications and side effects between LA and RFA
Tolerability evaluated by McGill Pain Questionnaire | 0 and 6 months
  Tolerability will be evaluated by McGill Pain Questionnaire, Melzack 1975, italian version
Quality of Life | 6 months and 1 year
  Quality of Life will be evaluated by SF-36 QoL questionnaire after 6 months and 1 year in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Cianni, Principal Investigator — Santa Maria Goretti Hospital
Locations (1):
- Santa Maria Goretti Hospital, Latina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gharib H, Papini E, Paschke R, Duick DS, Valcavi R, Hegedus L, Vitti P; AACE/AME/ETA Task Force on Thyroid Nodules. American Association of Clinical Endocrinologists, Associazione Medici Endocrinologi, and European Thyroid Association medical guidelines for clinical practice for the diagnosis and management of thyroid nodules: executive summary of recommendations. J Endocrinol Invest. 2010;33(5 Suppl):51-6. PMID 20543551
- [Background] Pacella CM, Bizzarri G, Guglielmi R, Anelli V, Bianchini A, Crescenzi A, Pacella S, Papini E. Thyroid tissue: US-guided percutaneous interstitial laser ablation-a feasibility study. Radiology. 2000 Dec;217(3):673-7. doi: 10.1148/radiology.217.3.r00dc09673. PMID 11110927
- [Background] Ahmed M, Brace CL, Lee FT Jr, Goldberg SN. Principles of and advances in percutaneous ablation. Radiology. 2011 Feb;258(2):351-69. doi: 10.1148/radiol.10081634. PMID 21273519
- [Background] Papini E, Guglielmi R, Bizzarri G, Graziano F, Bianchini A, Brufani C, Pacella S, Valle D, Pacella CM. Treatment of benign cold thyroid nodules: a randomized clinical trial of percutaneous laser ablation versus levothyroxine therapy or follow-up. Thyroid. 2007 Mar;17(3):229-35. doi: 10.1089/thy.2006.0204. PMID 17381356
- [Background] Cesareo R, Pasqualini V, Simeoni C, Sacchi M, Saralli E, Campagna G, Cianni R. Prospective study of effectiveness of ultrasound-guided radiofrequency ablation versus control group in patients affected by benign thyroid nodules. J Clin Endocrinol Metab. 2015 Feb;100(2):460-6. doi: 10.1210/jc.2014-2186. Epub 2014 Nov 11. PMID 25387256